CLINICAL TRIAL: NCT01543503
Title: A Global Comparative Observational Study In Rheumatoid Arthritis (RA) Patients Who Are Treated With A TNF Inhibitor Or Tocilizumab As The First Biologic Therapy
Brief Title: An Global Comparative Observational Study of RoActemra/Actemra (Tocilizumab) in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MA27950
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Results first posted 2016-02-10 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective, multi-center, observational study will assess the efficacy and safety of treatment in patients who are treated with a TNF Inhibitor or RoActemra/Actemra (tocilizumab) as the first biologic therapy. Data will be collected for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Diagnosis of rheumatoid arthritis
* Non-respondent or intolerant to non-biologic disease-modifying anti-rheumatic drug (DMARD) therapy
* Patient has been prescribed a first biologic therapy up to 6 weeks prior to the inclusion visit, irrespective of the treatment prescribed

Exclusion Criteria:

* Patients whose first biologic therapy is given as part of a clinical trial studying rheumatoid arthritis (RA) treatment
* Patients who are receiving or have received experimental DMARDs as part of a clinical trial studying RA treatment in the last 12 months
* Patients whose first biologic is rituximab, abatacept or anakinra.
* Patients who have received any biologic therapy for more than 6 weeks prior to the inclusion visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with rheumatoid arthritis
Sampling Method: Probability Sample
Enrollment: 1225 (Actual)
Dates: Start 2012-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (131):
- Argentina (3):
  - Catamarca Capital
  - Mendoza
  - Rosario
- Belgium (13):
  - Aalst
  - Assebroek
  - Aye
  - Brussels
  - Edegem
  - Genk
  - Ghent
  - Godinne
  - Heusy
  - Liège
  - Ostend
  - Verviers
  - Westmalle
- Colombia (4):
  - Barranquilla
  - Bogotá
  - Bucaramanga
  - Medellín
- Ecuador (5):
  - Cuenca
  - Esmeraldas
  - Guayaquil
  - Portoviejo
  - Quito
- Germany (20):
  - Aachen
  - Bad Aibling
  - Bad Neuenahr-Ahrweiler
  - Bayreuth
  - Berlin
  - Cologne
  - Dresden
  - Erfurt
  - Erlangen
  - Fulda
  - Hamburg
  - Heidelberg
  - Herne
  - Ludwigsfelde
  - München
  - Passau
  - Rostock
  - Stuttgart
  - Traunstein
  - Wuppertal
- Greece (3):
  - Athens
  - Pátrai
  - Thessaloniki
- Guatemala City, Guatemala
- Italy (21):
  - Coppito, Abruzzo
  - Pescara, Abruzzo
  - Brindisi, Apulia
  - Martina Franca, Apulia
  - San Cesario di Lecce, Apulia
  - Reggio Calabria, Calabria
  - Avellino, Campania
  - Napoli, Campania
  - Salerno, Campania
  - Udine, Friuli Venezia Giulia
  - Rome, Lazio
  - Arenzano, Liguria
  - Brescia, Lombardy
  - Legnano, Lombardy
  - Milan, Lombardy
  - Agnone, Molise
  - Turin, Piedmont
  - Catania, Sicily
  - Jesi Ancona, The Marches
  - Prato, Tuscany
  - Perugia, Umbria
- Mexico (3):
  - Guadalajara
  - Mexicali
  - Mexico Ctiy
- Panama City, Panama
- Portugal (5):
  - Almada
  - Amadora
  - Lisbon
  - Porto
  - Vila Nova de Gaia
- Spain (3):
  - Fuenlabrada, Madrid
  - Madrid, Madrid
  - San Sebastián de los Reyes, Madrid
- Switzerland (4):
  - Aarau
  - Basel
  - Chur
  - Sankt Gallen
- Ukraine (7):
  - Donetsk
  - Kharkiv
  - Kmelnytskyy
  - Kyiv
  - Odesa
  - Uzhhorod
  - Zaporizhzhya
- United Kingdom (37):
  - Barnsley
  - Basildon
  - Basingstoke
  - Brighton
  - Cannock
  - Cardiff
  - Chertsey
  - Crawley
  - Darlington
  - Enfield
  - Grimsby
  - Guildford
  - Ipswich
  - Kettering
  - Lancaster
  - Leeds
  - Llandudno
  - London
  - Luton
  - Maidstone
  - Margate
  - Metropolitan Borough of Wirral
  - North Shields
  - Oswestry
  - Plymouth
  - Portsmouth
  - Reading
  - Rhyl
  - Romford
  - Sheffield
  - Stockport
  - Sunderland
  - Swindon
  - Torquay
  - Warrington
  - Wolverhampton
  - Wrightington
- Montevideo, Uruguay

REFERENCES:
- [Derived] Choy EH, Bernasconi C, Aassi M, Molina JF, Epis OM. Treatment of Rheumatoid Arthritis With Anti-Tumor Necrosis Factor or Tocilizumab Therapy as First Biologic Agent in a Global Comparative Observational Study. Arthritis Care Res (Hoboken). 2017 Oct;69(10):1484-1494. doi: 10.1002/acr.23303. Epub 2017 Sep 6. PMID 28622454

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This observational study was conducted at 158 sites in 16 countries from 9 February 2012 to 20 February 2015.
Pre-assignment Details: A total of 1250 participants were screened for entry into the study, with 1225 participants enrolled in the study. One participant whose randomization status was unknown withdrew informed consent.
Groups:
- Tocilizumab: Participants with rheumatoid arthritis who were currently being treated with tocilizumab as a first biologic therapy and were non-responders or intolerant to conventional synthetic disease-modifying anti-rheumatic drug (csDMARD) therapy. Tocilizumab administration occurred as per routine practice and following the local prescribing information. Participants were observed for 52 weeks after initiation of the first biologic therapy. Participants who stopped treatment with the prescribed tocilizumab for reasons of inefficacy or intolerance continued to be observed for the planned period of 52 weeks.
- TNF Inhibitor: Participants with rheumatoid arthritis who were currently being treated with a TNF inhibitor as a first biologic therapy and were non-responders or intolerant to csDMARD therapy. The TNF inhibitor administration occurred as per routine practice and following the local prescribing information. Participants were observed for 52 weeks after initiation of the first biologic therapy. Participants who stopped treatment with the prescribed TNF inhibitor for reasons of inefficacy or intolerance continued to be observed for the planned period of 52 weeks.
Period: Overall Study
Arm/Group | Tocilizumab | TNF Inhibitor
Started | 426 | 798
Completed | 350 | 711
Not Completed | 76 | 87
Not completed — Lost to Follow-up | 32 | 36
Not completed — Adverse Event | 9 | 13
Not completed — Lack of Efficacy | 4 | 16
Not completed — Participant withdrew informed consent | 8 | 10
Not completed — Change of jobs | 0 | 1
Not completed — Intolerance to the biologic treatment | 0 | 1
Not completed — Probable overlap of RA with fibromyalgia | 1 | 0
Not completed — Participant did not complete last visit | 0 | 2
Not completed — Refused to continue treatment | 7 | 0
Not completed — Incorrect medication received | 1 | 0
Not completed — Participant moved to another city | 2 | 0
Not completed — Participant will not return for visits | 0 | 2
Not completed — Participant transferred to another city | 1 | 0
Not completed — Participant moved to Scotland | 1 | 0
Not completed — Participant decision to stop treatment | 1 | 0
Not completed — Investigator did not wish to participate | 1 | 1
Not completed — Participant recruited after closing date | 0 | 1
Not completed — Site stopped participation | 5 | 1
Not completed — Participant did not attend a visit | 1 | 0
Not completed — Moved to other rheumatologic site | 0 | 1
Not completed — Participant consented to another study | 0 | 2
Not completed — Participant went to United States | 1 | 0
Not completed — Screen failure | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were described for the safety population. All enrolled participants who received at least one dose of a TNF inhibitor or tocilizumab during the study were included in the safety population.
Groups:
- Tocilizumab: Participants with rheumatoid arthritis who were currently being treated with tocilizumab as a first biologic therapy and were non-responders or intolerant to csDMARD therapy. Tocilizumab administration occurred as per routine practice and following the local prescribing information. Participants were observed for 52 weeks after initiation of the first biologic therapy. Participants who stopped treatment with the prescribed tocilizumab for reasons of inefficacy or intolerance continued to be observed for the planned period of 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Tocilizumab | TNF Inhibitor | Total
Number analyzed (Participants) | 423 | 793 | 1216
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.26 (12.75) | 55.16 (13.05) | 54.85 (12.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 351 | 615 | 966
  Male | 72 | 178 | 250

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Calculated Disease Activity Score Based on 28 Joint Count Erythrocyte Sedimentation Rate at Week 24
Description: Disease activity score based on 28 joint counts (DAS28) is a composite measure of disease severity and it incorporates four specific measures of disease: swollen joint count (SJC) of 28 joints, tender joint count (TJC) of 28 joints, Patient's Global Assessment of Disease Activity by visual analogue scale (VAS), and acute-phase inflammatory marker [erythrocyte sedimentation rate (ESR) in millimeter/hour (mm/h), or C-reactive protein (CRP) in milligram/liter (mg/L)]. For the purposes of this study, ESR was used whenever possible to calculate the DAS28 (DAS28-ESR). Higher the scores, greater is the disease activity. A DAS28 score of less than or equal to (</=) 3.2 = low disease activity, a DAS28 score of >3.2 to 5.1 = moderate to high disease activity.
Time Frame: Baseline and Week 24
Population: Participants belonging to the safety population who had first biologic administration within 60 days after the last Rheumatoid Arthritis (RA) disease activity assessment were included in the effectiveness analysis population. Data of participants available at the time of the assessment were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 155 | 314
Units on a scale | -2.795 [-3.107 to -2.483] | -1.945 [-2.249 to -1.640]
Statistical Analysis 1: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor: Analysis is based on an analysis of covariance (ANCOVA) model with change from baseline in DAS28-ESR at 24 weeks as dependent variable; therapy, site country, and treatment as fixed effects; DAS28-ESR at baseline as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -0.851, 95% CI 2-sided [-1.112 to -0.589]

2. Secondary Outcome: Mean Change From Baseline in Disease Activity Score Based on 28 Joint Count Erythrocyte Sedimentation Rate at Week 52
Description: Disease activity score based on 28 joint counts (DAS28) is a composite measure of disease severity and it incorporates four specific measures of disease: swollen joint count (SJC) of 28 joints, tender joint count (TJC) of 28 joints, Patient's Global Assessment of Disease Activity by visual analogue scale (VAS), and acute-phase inflammatory marker (ESR in mm/h, or CRP in mg/L). For the purposes of this study, ESR was used whenever possible to calculate the DAS28 (DAS28-ESR). Higher the scores, greater is the disease activity. A DAS28 score of </= 3.2 = low disease activity, a DAS28 score of >3.2 to 5.1 = moderate to high disease activity.
Time Frame: Baseline and Week 52
Population: The effectiveness analysis population was used for analysis. Data of participants available at the time of the assessment were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 142 | 282
units on a scale | -3.015 [-3.279 to -2.751] | -2.105 [-2.325 to -1.885]
Statistical Analysis 1: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor: Analysis is based on an ANCOVA model with change from baseline to 12 months in DAS28-ESR as dependent variable; therapy and treatment as fixed effects; DAS28-ESR at baseline as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -0.910, 95% CI 2-sided [-1.204 to -0.617]

3. Secondary Outcome: Mean Change From Baseline in Erythrocyte Sedimentation Rate
Description: Blood samples were collected for ESR, which is an acute phase reactant and a measure of inflammation. BL = baseline.
Time Frame: Baseline, Week 24, Week 52
Population: The effectiveness analysis population was used for analysis. n = the number of participants available for assessment at a given time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm/hr
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 390 | 693
mm/hr
  Change from BL to Week 24, n = 225, 456 | -22.732 [-24.717 to -20.747] | -9.502 [-11.112 to -7.892]
  Change from BL to Week 52, n = 215, 411 | -21.515 [-23.875 to -19.155] | -8.868 [-10.865 to -6.870]
Statistical Analysis 1: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor for ESR at Week 24: Analysis is based on an ANCOVA model with change from baseline to 6 months in ESR as a dependent variable; therapy and treatment as fixed effects; ESR at baseline as the covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -13.230, 95% CI 2-sided [-15.513 to -10.947]
Statistical Analysis 2: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor for ESR at Week 52: Analysis is based on an ANCOVA model with change from baseline to 12 months in ESR, as the dependent variable; therapy and treatment as fixed effects; ESR at baseline as the covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -12.648, 95% CI 2-sided [-15.419 to -9.876]

4. Secondary Outcome: Mean Change From Baseline in C-reactive Protein
Description: Blood samples were collected for C-reactive protein (CRP). CRP is an inflammation marker. High levels of this protein indicate inflammation in diseases such as RA.
Time Frame: Baseline, Week 24, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 390 | 693
mg/L
  Change from BL to Week 24, n = 177, 396 | -11.005 [-14.131 to -7.880] | -4.333 [-6.859 to -1.807]
  Change from BL to Week 52, n = 173, 348 | -6.332 [-10.524 to -2.140] | -5.216 [-8.711 to -1.722]
Statistical Analysis 1: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor for CRP at Week 24: Analysis is based on an ANCOVA model with change from baseline to 6 months in CRP as a dependent variable; therapy and treatment as fixed effects; CRP at baseline as the covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -6.673, 95% CI 2-sided [-10.271 to -3.074]
Statistical Analysis 2: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor for CRP at Week 52: Analysis is based on an ANCOVA model with change from baseline to 12 months in CRP as the dependent variable; therapy and treatment as fixed effects; CRP at baseline as the covariate; Test type: Superiority or Other; p = 0.659, ANCOVA; Mean Difference (Net) = -1.116, 95% CI 2-sided [-6.074 to 3.842]

5. Secondary Outcome: Mean Change From Baseline in Swollen Joint Count
Description: A swollen joint count (SJC) is the most specific clinical method to quantify abnormalities in participants with RA. It reflects the amount of inflamed synovial tissue. Twenty-eight joints were assessed for swelling. Joints were classified as swollen (1)/ not swollen (0) giving a total possible SJC score of 0 to 28.
Time Frame: Baseline, Week 24, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of swollen joints
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 390 | 693
Number of swollen joints
  Change from BL to Week 24, n = 288, 554 | -5.698 [-6.124 to -5.273] | -5.122 [-5.480 to -4.764]
  Change from BL to Week 52, n = 258, 503 | -6.313 [-6.724 to -5.902] | -5.561 [-5.909 to -5.213]
Statistical Analysis 1: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor for SJC at Week 24: Analysis is based on an ANCOVA model with change from baseline to 6 months in SJC as the dependent variable; therapy and treatment as fixed effects; SJC at baseline as the covariate; Test type: Superiority or Other; p = 0.024, ANCOVA; Mean Difference (Net) = -0.576, 95% CI 2-sided [-1.078 to -0.075]
Statistical Analysis 2: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor for SJC at Week 52: Analysis is based on an ANCOVA model with change from baseline to 12 months in SJC, as the dependent variable; therapy and treatment as fixed effects; SJC, at baseline as the covariate; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Net) = -0.752, 95% CI 2-sided [-1.238 to -0.267]

6. Secondary Outcome: Mean Change From Baseline in Tender Joint Count
Description: A tender joint count (TJC) is the most specific clinical method to quantify abnormalities in participants with RA. It is associated with the level of pain. Twenty-eight joints were assessed for tenderness. Joints were classified as tender (1)/not tender (0) giving a total possible TJC score of 0 to 28.
Time Frame: Baseline, Week 24, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of tender joints
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 390 | 693
Number of tender joints
  Change from BL to Week 24, n = 289, 554 | -7.922 [-8.593 to -7.251] | -7.302 [-7.868 to -6.736]
  Change from BL to Week 52, n = 259, 501 | -8.421 [-9.122 to -7.720] | -7.205 [-7.799 to -6.610]
Statistical Analysis 1: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor for TJC at Week 24: Analysis is based on an ANCOVA model with change from baseline to 6 months in TJC as the dependent variable; therapy and treatment as fixed effects; TJC at baseline as the covariate; Test type: Superiority or Other; p = 0.123, ANCOVA; Mean Difference (Net) = -0.620, 95% CI 2-sided [-1.408 to 0.169]
Statistical Analysis 2: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor for TJC at Week 52: Analysis is based on an ANCOVA model with change from baseline to 12 months in TJC as the dependent variable; therapy and treatment as fixed effects; TJC at baseline as the covariate; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Net) = -1.216, 95% CI 2-sided [-2.039 to -0.393]

7. Secondary Outcome: Mean Change From Baseline in Clinical Disease Activity Index and Simplified Disease Activity Index Score
Description: Clinical Disease Activity Index (CDAI) was calculated as the sum of the following parameters: SJC + TJC + VAS Patient Global Assessment of Disease Activity + VAS Physician Global Assessment of Disease Activity. VAS assessments involved a 10-cm horizontal scale from 'no disease activity' to 'maximum disease activity'. CDAI scores ranged from 0 to 76, with higher scores indicating increased disease activity. Simplified Disease Activity Index (SDAI) was calculated as the sum of the following parameters: SJC +TJC + Patient Global Assessment of Disease Activity + Physician Global Assessment of Disease Activity + CRP. SDAI scores ranged from 0 to 86, with higher scores also indicating increased disease activity.
Time Frame: Baseline, Week 24, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 390 | 693
units on a scale
  CDAI, Change from BL to Week 24, n = 176, 286 | -20.251 [-21.934 to -18.568] | -16.776 [-18.280 to -15.271]
  CDAI, Change from BL to Week 52, n = 162, 267 | -22.846 [-24.634 to -21.058] | -18.246 [-19.823 to -16.669]
  SDAI, Change from BL to Week 24, n = 93, 193 | -21.394 [-23.668 to -19.120] | -18.164 [-20.051 to -16.278]
  SDAI, Change from BL to Week 52, n = 91, 169 | -22.294 [-24.791 to -19.797] | -19.048 [-21.128 to -16.969]
Statistical Analysis 1: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor for CDAI score at Week 24: Analysis is based on an ANCOVA model with change from baseline to 6 months in CDAI the dependent variable; therapy and treatment as fixed effects; CDAI at baseline as the covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -3.475, 95% CI 2-sided [-5.481 to -1.469]
Statistical Analysis 2: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor for CDAI score at Week 52: Analysis is based on an ANCOVA model with change from baseline to 12 months in CDAI as the dependent variable; therapy and treatment as fixed effects; CDAI at baseline as the covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -4.600, 95% CI 2-sided [-6.708 to -2.492]
Statistical Analysis 3: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor for SDAI score at Week 24: Analysis is based on an ANCOVA model with change from baseline to 6 months in SDAI as the dependent variable; therapy and treatment as fixed effects; SDAI at baseline as the covariate; Test type: Superiority or Other; p = 0.014, ANCOVA; Mean Difference (Net) = -3.229, 95% CI 2-sided [-5.806 to -0.652]
Statistical Analysis 4: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor for SDAI score at Week 52: Analysis is based on an ANCOVA model with change from baseline to 12 months in SDAI as the dependent variable; therapy and treatment as fixed effects; SDAI at baseline as the covariate; Test type: Superiority or Other; p = 0.027, ANCOVA; Mean Difference (Net) = -3.245, 95% CI 2-sided [-6.121 to -0.370]

8. Secondary Outcome: Mean Change From Baseline in Physician Global Assessment Score
Description: The Physician's Global Assessment of disease activity was assessed using a 0 to 100 millimeter (mm) horizontal VAS. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). Change from baseline = scores at observation minus score at baseline. An increase in score from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline, Week 24, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 390 | 693
scores on a scale
  Change from BL to Week 24, n = 183, 300 | -35.581 [-38.656 to -32.506] | -26.551 [-29.293 to -23.809]
  Change from BL to Week 52, n = 174, 287 | -37.359 [-40.631 to -34.087] | -27.122 [-30.042 to -24.202]
Statistical Analysis 1: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor for Physician Global Assessment score at Week 24: Analysis is based on an ANCOVA model with change from baseline to 6 months in Physician Global Assessment of Disease Activity as the dependent variable; therapy and treatment as fixed effects; Physician Global Assessment of Disease Activity at baseline as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -9.030, 95% CI 2-sided [-12.655 to -5.404]
Statistical Analysis 2: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor for Physician Global Assessment score at Week 52: Analysis is based on an ANCOVA model with change from baseline to 12 months in Physician Global Assessment of Disease Activity as the dependent variable; therapy and treatment as fixed effects; Physician Global Assessment of Disease Activity at baseline as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -10.237, 95% CI 2-sided [-14.130 to -6.345]

9. Secondary Outcome: Loss of Efficacy or Development of Intolerance to Biologic Therapy
Description: Events that are clearly consistent with the expected pattern of progression of the underlying disease may contribute to lack of efficacy. Lack of efficacy was one of the reasons for termination of biology therapy. The number of participants showing lack of efficacy to biologic therapy is presented.
Time Frame: Up to Week 52
Population: The safety population included all recruited participants who received at least one dose of a TNF inhibitor or tocilizumab during the study.
Measure: Number; unit: participants
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 423 | 793
participants | 15 | 106

10. Secondary Outcome: Proportion of Participants Who Terminated Biologic Treatment
Description: The proportion of participants who discontinued biologic treatment was compared between tocilizumab-treated and TNF inhibitor-treated participants.
Time Frame: Up to Week 52
Population: The safety population was used for analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 423 | 793
Percentage of participants | 14.9 | 27.4

11. Secondary Outcome: Reasons for Treatment Discontinuation
Description: The reasons for discontinuation of tocilizumab or TNF inhibitor is presented.
Time Frame: Up to Week 52
Population: The safety population was used for analysis.
Measure: Number; unit: participants
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 423 | 793
participants
  Adverse event | 24 | 87
  Lack of efficacy | 15 | 106
  Other | 24 | 23

12. Secondary Outcome: Cumulative Number of Participants Who Discontinued Biologic Therapy at the End of Each Study Period
Description: The total number of participants who discontinued biologic therapy at the end of each study period (Week 0 - 24, Week 24 - 52, Week 52 - 57 and Week 57 - end of treatment) is presented. Participants who did not have a biologic therapy discontinuation or discontinued before having one, were considered as 'censored' at the date study termination.
Time Frame: Up to end of treatment
Population: The safety population was used for analysis.
Measure: Number; unit: participants
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 423 | 793
participants
  Week 0 -24 | 36 | 119
  Week 24 - 52 | 61 | 208
  Week 52 - 57 | 62 | 212
  Week 57 - End of treatment | 63 | 216
Statistical Analysis 1: Comparison: Tocilizumab vs TNF Inhibitor; Test type: Superiority or Other; p < 0.001, Log Rank

13. Secondary Outcome: Number of Participants of Infusion Reactions or Injection Site Reactions During the Study Following the Start of the First Biologic Therapy
Description: An infusion reaction was defined as an adverse event (AE) occurring during and within 24 hours after the infusion, which may include hypersensitivity reactions or anaphylactic reactions. Injection site reactions were included in the summaries for infusion reactions.
Time Frame: Up to Week 52
Population: The safety population was used for analysis.
Measure: Number; unit: participants
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 423 | 793
participants
  Participants with Non-Serious infusion reaction | 33 | 75
  Participants with Serious infusion reaction | 4 | 3

14. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Non-serious Adverse Events
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to Week 52
Population: The safety population was used for analysis.
Measure: Number; unit: participants
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 423 | 793
participants
  Participants with AE | 208 | 449
  Participants with SAE | 22 | 64
  Participants with non-serious AE | 196 | 421

15. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events of Special Interest, Including Infections, During the Study
Description: Adverse events of special interest (AESI) for this study included: infections (including opportunistic infections), myocardial infarction/acute coronary syndrome, gastrointestinal perforation and related events, malignancies, anaphylaxis / hypersensitivity reactions, demyelinating disorders, stroke, bleeding events and hepatic events. Based on seriousness criteria, they were categorized as serious and non-serious adverse events of special interest.
Time Frame: Up to Week 52
Population: The safety population was used for analysis.
Measure: Number; unit: participants
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 423 | 793
participants
  Participants with Serious AESI | 13 | 27
  Participants with Non-Serious AESI | 22 | 16

16. Secondary Outcome: Mean Change From Baseline in Health Assessment Questionnaire Disability Index Score
Description: The Health Assessment Questionnaire-Disability Index (HAQ-DI) is a 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping and activities of daily living). Responses in each functional area are scored from 0 to 3 (0=no difficulty and 3=inability to perform a task in that area). HAQ-DI total scores expressed as overall mean score with range 0-3: 0-0.25=normal functioning; 0.25-0.5=mild functional limitation; 0.5-1=moderate functional limitation; more than 1=significant functional limitation.
Time Frame: Baseline, Week 24, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 390 | 693
Scores on a scale
  Change from BL to Week 24, n = 169, 301 | -0.591 [-0.694 to -0.488] | -0.445 [-0.538 to -0.352]
  Change from BL to Week 52, n = 152, 255 | -0.593 [-0.710 to -0.476] | -0.430 [-0.539 to -0.320]
Statistical Analysis 1: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor at Week 24: Analysis is based on an ANCOVA model with change from baseline to 6 months in HAQ-DI as dependent variable; therapy and treatment as fixed effects; HAQ-DI at baseline as covariates; Test type: Superiority or Other; p = 0.020, ANCOVA; Mean Difference (Net) = -0.146, 95% CI 2-sided [-0.269 to -0.024]
Statistical Analysis 2: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor at Week 52: Analysis is based on an ANCOVA model with change from baseline to 12 months in HAQ-DI as dependent variable; therapy and treatment as fixed effects; HAQ-DI at baseline as covariates; Test type: Superiority or Other; p = 0.020, ANCOVA; Mean Difference (Net) = -0.164, 95% CI 2-sided [-0.301 to -0.026]

17. Secondary Outcome: Mean Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue Score
Description: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the participant's fatigue. The sum of all responses resulted in the FACIT-F score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflects an improvement in the participant's health status.
Time Frame: Baseline, Week 24, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 390 | 693
scores on a scale
  Change from BL to Week 24, n = 64, 86 | -7.153 [-10.003 to -4.304] | -3.260 [-6.279 to -0.242]
  Change from BL to Week 52, n = 50, 77 | -4.566 [-7.822 to -1.310] | -1.779 [-5.096 to 1.538]
Statistical Analysis 1: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor at Week 24: Analysis is based on an ANCOVA model with change from baseline to 6 months in FACIT-F score as dependent variable; therapy and treatment as fixed effects; FACIT-F score at baseline as covariates; Test type: Superiority or Other; p = 0.032, ANCOVA; Mean Difference (Net) = -3.893, 95% CI 2-sided [-7.457 to -0.329]
Statistical Analysis 2: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor for Week 52: Analysis is based on an ANCOVA model with change from baseline to 12 months in FACIT-F score as dependent variable; therapy and treatment as fixed effects; FACIT-F score at baseline as covariates; Test type: Superiority or Other; p = 0.168, ANCOVA; Mean Difference (Net) = -2.787, 95% CI 2-sided [-6.763 to 1.189]

18. Secondary Outcome: Mean Change From Baseline in Visual Analogue Scale Pain Score
Description: VAS is a 100 mm scale. Intensity of pain range: 0 mm=no pain to 100 mm=worst possible pain. Change from baseline =scores at observation minus score at baseline. An increase in score from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline, Week 24, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 390 | 693
units on a scale
  Change from BL to Week 24, n = 204, 378 | -29.308 [-32.922 to -25.694] | -23.647 [-26.664 to -20.630]
  Change from BL to Week 52, n = 183, 336 | -32.957 [-36.711 to -29.202] | -23.155 [-26.386 to -19.923]
Statistical Analysis 1: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor at Week 24: Analysis is based on an ANCOVA model with change from baseline to 6 months in participant's VAS score as dependent variable; therapy and treatment as fixed effects; participant's VAS score at baseline as covariates; Test type: Superiority or Other; p = 0.009, ANCOVA; Mean Difference (Net) = -5.661, 95% CI 2-sided [-9.912 to -1.411]
Statistical Analysis 2: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor at Week 52: Analysis is based on an ANCOVA model with change from baseline to 12 months in participant's VAS score as dependent variable; therapy and treatment as fixed effects; participant's VAS score at baseline as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -9.802, 95% CI 2-sided [-14.245 to -5.360]

19. Secondary Outcome: Shift From Baseline in Morning Stiffness
Description: Shift tables presenting the number of participants in each bivariate category Week (W) 0 versus Week 24 and Week 52, with regards to morning stiffness at the different time points, was presented for each treatment arm. For participants who experienced joint stiffness while waking up in the morning, duration of morning stiffness was categorized as follows: Less than 30 minutes (min), Between 30 and 60 minutes, Between 60 and 120 minutes, Between 120 to 240 minutes, More than 240 minutes and the whole day. Baseline = BL
Time Frame: Baseline, Week 24, Week 52
Population: The effectiveness analysis population was used for analysis.
Measure: Number; unit: participants
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 390 | 693
participants
  BL, < 30 min; W 24, < 30 min | 13 | 19
  BL, < 30 min; W 24, 30-60 min | 1 | 8
  BL, < 30 min; W 24, 60-120 min | 2 | 1
  BL, < 30 min; W 24, 120-240 min | 0 | 1
  BL, < 30 min; W 24, > 240 min | 0 | 0
  BL, < 30 min; W 24, the whole day | 1 | 0
  BL, between 30-60 min; W 24 < 30 min | 19 | 49
  BL, between 30-60 min; W 24, 30-60 min | 9 | 30
  BL, between 30-60 min; W 24, 60-120 min | 1 | 3
  BL, between 30-60 min; W 24, 120-240 min | 0 | 1
  BL, between 30-60 min; W 24, > 240 min | 0 | 0
  BL, between 30-60 min; W 24, the whole day | 0 | 0
  BL, between 60-120 min; W 24, < 30 min | 22 | 34
  BL, between 60-120 min; W 24, 30-60 min | 17 | 22
  BL, between 60-120 min; W 24, 60-120 min | 4 | 7
  BL, between 60-120 min; W 24, 120-240 min | 0 | 0
  BL, between 60-120 min; W 24, > 240 min | 0 | 0
  BL, between 60-120 min; W 24, the whole day | 0 | 1
  BL, between 120-240 min; W 24, < 30 min | 12 | 10
  BL, between 120-240 min; W 24, 30-60 min | 6 | 9
  BL, between 120-240 min; W 24, 60-120 min | 2 | 8
  BL, between 120-240 min; W 24, 120-240 min | 3 | 4
  BL, between 120-240 min; W 24, > 240 min | 0 | 1
  BL, between 120-240 min; W 24, the whole day | 0 | 0
  BL, more than 240 min; W 24, < 30 min | 0 | 7
  BL, more than 240 min; W 24, 30-60 min | 2 | 2
  BL, more than 240 min; W 24, 60-120 min | 0 | 0
  BL, more than 240 min; W 24, 120-240 min | 0 | 0
  BL, more than 240 min; W 24, > 240 min | 0 | 1
  BL, more than 240 min; W 24, the whole day | 0 | 0
  BL, the whole day; W 24, < 30 min | 1 | 2
  BL, the whole day; W 24, 30-60 min | 3 | 2
  BL, the whole day; W 24, 60-120 min | 2 | 5
  BL, the whole day; W 24, 120-240 min | 0 | 1
  BL, the whole day; W 24, > 240 min | 0 | 0
  BL, the whole day; W 24, the whole day | 1 | 1
  BL, < 30 min; W 52, < 30 min | 6 | 13
  BL, < 30 min; W 52, 30-60 min | 2 | 4
  BL, < 30 min; W 52, 60-120 min | 0 | 0
  BL, < 30 min; W 52, 120-240 min | 2 | 1
  BL, < 30 min; W 52, > 240 min | 0 | 1
  BL, < 30 min; W 52, the whole day | 0 | 0
  BL, between 30-60 min; W 52, < 30 min | 17 | 43
  BL, between 30-60 min; W 52, 30-60 min | 9 | 19
  BL, between 30-60 min; W 52, 60-120 min | 1 | 5
  BL, between 30-60 min; W 52, 120-240 min | 0 | 1
  BL, between 30-60 min; W 52, > 240 min | 0 | 0
  BL, between 30-60 min; W 52, the whole day | 0 | 0
  BL, between 60-120 min; W 52, < 30 min | 20 | 33
  BL, between 60-120 min; W 52, 30-60 min | 8 | 21
  BL, between 60-120 min; W 52, 60-120 min | 4 | 4
  BL, between 60-120 min; W 52, 120-240 min | 0 | 3
  BL, between 60-120 min; W 52, > 240 min | 0 | 2
  BL, between 60-120 min; W 52, the whole day | 1 | 0
  BL, between 120-240 min; W 52, < 30 min | 14 | 9
  BL, between 120-240 min; W 52, 30-60 min | 6 | 6
  BL, between 120-240 min; W 52, 60-120 min | 5 | 8
  BL, between 120-240 min; W 52, 120-240 min | 1 | 3
  BL, between 120-240 min; W 52, > 240 min | 0 | 1
  BL, between 120-240 min; W 52, the whole day | 0 | 1
  BL, more than 240 min; W 52, < 30 min | 0 | 5
  BL, more than 240 min; W 52, 30-60 min | 2 | 4
  BL, more than 240 min; W 52, 60-120 min | 0 | 0
  BL, more than 240 min; W 52, 120-240 min | 1 | 0
  BL, more than 240 min; W 52, > 240 min | 0 | 0
  BL, more than 240 min; W 52, the whole day | 0 | 1
  BL, the whole day; W 52, < 30 min | 2 | 3
  BL, the whole day; W 52, 30-60 min | 1 | 2
  BL, the whole day; W 52, 60-120 min | 2 | 2
  BL, the whole day; W 52, 120-240 min | 0 | 1
  BL, the whole day; W 52, > 240 min | 0 | 0
  BL, the whole day; W 52, the whole day | 0 | 0

20. Secondary Outcome: Change From Baseline in Patient Global Assessment of Disease Activity
Description: The patient's global assessment of disease activity is assessed on a 0 to 100 mm horizontal VAS by the participant. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 24, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Tocilizumab | TNF Inhibitor
Number analyzed (Participants) | 390 | 693
scores on a scale
  Change from BL to Week 24, n = 225, 423 | -29.633 [-32.994 to -26.273] | -24.525 [-27.388 to -21.662]
  Change from BL to Week 52, n = 206, 378 | -31.919 [-35.630 to -28.209] | -24.153 [-27.385 to -20.921]
Statistical Analysis 1: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor at Week 24: Analysis is based on an ANCOVA model with change from baseline to 6 months in Patient's Global Assessment of Disease as dependent variable; therapy and treatment as fixed effects; Patient's Global Assessment of Disease at baseline as covariates; Test type: Superiority or Other; p = 0.010, ANCOVA; Mean Difference (Net) = -5.108, 95% CI 2-sided [-9.017 to -1.200]
Statistical Analysis 2: Comparison: Tocilizumab vs TNF Inhibitor; Treatment Difference between Tocilizumab and TNF inhibitor at Week 52: Analysis is based on an ANCOVA model with change from baseline to 12 months in Patient's Global Assessment of Disease as dependent variable; therapy and treatment as fixed effects; Patient's Global Assessment of Disease at baseline as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -7.767, 95% CI 2-sided [-12.161 to -3.372]

ADVERSE EVENTS:
Time Frame: Up to Week 52
Description: SAEs and non-serious AEs were reported for members of the safety population, which included all recruited participants who received at least one dose of a TNF inhibitor or tocilizumab during the study. All SAEs are reported, without any frequency threshold.
Arm/Group | Tocilizumab | TNF Inhibitor
Serious Adverse Events (participants affected / at risk) | 22/423 | 64/793
Other Adverse Events (participants affected / at risk) | 132/423 | 231/793
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=423) | TNF Inhibitor (N=793)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Parophthalmia (Eye disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Chest pain (General disorders) | 0 | 3
Injection site rash (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Ulcer (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 2
Abscess (Infections and infestations) | 0 | 1
Abscess of salivary gland (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cytomegalovirus gastritis (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2
Graft infection (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 6
Osteomyelitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 2 | 6
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 3
Staphylococcal infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Wound infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 3
Demyelination (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Depression (Psychiatric disorders) | 1 | 0
Glomerulonephritis membranous (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=423) | TNF Inhibitor (N=793)
NEUTROPENIA (Blood and lymphatic system disorders) | 14 | 3
DIARRHOEA (Gastrointestinal disorders) | 4 | 9
NAUSEA (Gastrointestinal disorders) | 9 | 15
INJECTION SITE REACTION (General disorders) | 1 | 22
BRONCHITIS (Infections and infestations) | 11 | 13
CELLULITIS (Infections and infestations) | 2 | 8
HERPES ZOSTER (Infections and infestations) | 4 | 8
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 15 | 35
NASOPHARYNGITIS (Infections and infestations) | 13 | 18
PHARYNGITIS (Infections and infestations) | 5 | 4
RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 | 10
SINUSITIS (Infections and infestations) | 6 | 8
URINARY TRACT INFECTION (Infections and infestations) | 15 | 26
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 8 | 13
NEUTROPHIL COUNT DECREASED (Investigations) | 5 | 8
TRANSAMINASES INCREASED (Investigations) | 10 | 4
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 9 | 5
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 10 | 7
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 11
HEADACHE (Nervous system disorders) | 7 | 23
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 | 12
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 9
ALOPECIA (Skin and subcutaneous tissue disorders) | 4 | 8
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 8
RASH (Skin and subcutaneous tissue disorders) | 9 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.